CLINICAL TRIAL: NCT04582279
Title: Application of Lung Ultrasound Artefact Analysis for Exclusion of Acute Rejection in Asymptomatic Lung Transplant Recipients
Brief Title: Lung Ultrasound Artefact Analysis for Exclusion of Acute Rejection in Lung Transplant Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tathagat Narula, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-002489
Record Dates: First submitted 2020-10-07; First posted 2020-10-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Post-Lung Transplantation Bronchiectasis
Keywords: Post lung transplant; Lung bronchoscopy; Lung biopsy; Lung rejection

STUDY DESIGN:
Intervention Model Description: There is only 1 group of participants being monitored. Every patient will follow the same study procedures
Masking Description: This study is not blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Receiving Ultrasound (Experimental): Every patient will receive a lung ultrasound prior to each scheduled bronchoscopy until the study stops.
  Interventions: Diagnostic Test: Lung ultrasound

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — The lung ultrasound will be performed by a trained pulmonologist by gently pressing a probe to various areas of your chest. This is a non-invasive procedure and you should not feel any pain. The ultrasound will take less than 10 minutes.

SUMMARY:
This study is being done to study a safe and non-invasive way to diagnose lung rejection and infection.

DETAILED DESCRIPTION:
Lung transplant recipients are at high risk for lung rejection and lung infection after transplant. This is diagnosed by performing lung bronchoscopies and lung biopsies. These procedures carry an increased risk for complications and are costly. This study is being done to study a safe and non-invasive way to diagnose lung rejection and infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 yrs) who had undergone single/double/heart-lung transplant
* Asymptomatic
* Normal spirometry defined as a FEV1 without significant drop from baseline (significant drop = >10% decrease from baseline)
* Clear chest radiograph over allograft

Exclusion Criteria:

* Patients who are unable to consent for the procedure
* Patients with subcutaneous emphysema or other technical challenges that could interfere with satisfactory image acquisition- as deemed by the operator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Establish predictive value of lung ultrasound | Month 0 to month 12
  Determine if lung ultrasound provides the same diagnostic results as bronchoscopy and biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Tathagat Narula, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials